CLINICAL TRIAL: NCT02697409
Title: Medical-student-delivered Smoking Prevention Program for Secondary Schools: The Education Against Tobacco Randomized Trial
Brief Title: Education Against Tobacco Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Giessen (Other)
Collaborators: University Hospital Tuebingen (Other); Universities of Giessen and Marburg Lung Center (Unknown)
Responsible Party: Principal Investigator, Titus J. Brinker, cand. med., University of Giessen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EATRCT
Record Dates: First submitted 2016-02-27; First posted 2016-03-03 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2016-05

CONDITIONS: Tobacco; Prevention; Adolescents; Schools

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): The intervention group receives two school-based modules taking less than two hours each delivered by medical students in the schools.
  Interventions: Behavioral: Education Against Tobacco intervention
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Education Against Tobacco intervention
  Arms: Intervention group

SUMMARY:
A two armed randomized trial is evaluating the effect of the medical-student-delivered school-based intervention Education Against Tobacco on the smoking behavior of adolescents in 7th grade of secondary school. The primary endpoint is the change in smoking prevalence between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Pupils of 7th grade of regular secondary schools in Germany

Exclusion Criteria:

* Not fulfilling the inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Smoking prevalence measured via questionnaire. | 24 months post baseline
  The difference in smoking prevalence at 24 months follow-up is the primary endpoint measured via questionnaires.

SECONDARY OUTCOMES:
Relevant differences due to the theory of planned behaviour between the two groups measured via questionnaire. | 24 months follow-up
  Difference in attitude towards smoking between the two groups at 24 months follow-up measured via questionnaires.
Changes in smoking behavior | 24 months post baseline
  The changes in smoking behavior (smoking onset, quitting) are studied as a secondary outcome measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Titus Brinker, Bünde, Germany

IPD SHARING:
Plan to Share IPD: Undecided